CLINICAL TRIAL: NCT03413332
Title: Web-Based Communication Education for Breast Cancer Survivorship Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Judy Wang, Associate Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-1407
Record Dates: First submitted 2018-01-05; First posted 2018-01-29 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: Chinese American Women; Provider-patient Communication; Survivorship Care
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-Talkcare Group (Experimental): use the web-based patient education tool
  Interventions: Other: E-Talkcare
- Usual Care Group (Placebo Comparator): receive usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: E-Talkcare — Women in the intervention group will receive the E-Talkcare web address, a user name, and a temporary password. The participant will be able to read or listen (through audio narration) to instructions on how to complete the intervention in order, though she can freely navigate between web modules. Each module will have an ever-present indicator (showing users' progress) and a link to for users to continue navigating through modules.We will ask participants to complete the full intervention within 3 months after intervention delivery and then complete a 3-month post-randomization interview (T1). The website will remain open for six months after intervention delivery to allow participants to use QPL if they wish. A 6-month post-randomization interview (T2) will then be administered.
  Arms: E-Talkcare Group
Other: Usual Care — Survivors randomized to the usual care group will receive care from their doctors as usual, allowing us to compare the intervention against real-world practice to inform next steps. Since we do not know if the intervention will be efficacious, we decided not to provide a delayed intervention to control participants.
  Arms: Usual Care Group

SUMMARY:
This two-phase research plan will develop and test a culturally relevant, web-based patient education program, hereafter known as E-Talkcare. The intervention aims to empower Chinese cancer patients to effectively communicate with different providers in different healthcare settings.

DETAILED DESCRIPTION:
This two-phase study develops and tests the usability and efficacy of a culturally relevant, web-based patient education program, hereafter known as E-Talkcare, in improving Chinese immigrant breast cancer survivors' competence, perceived control, and self-efficacy in cancer care communication (intermediate outcomes), and patient-reported symptoms, adherence to breast cancer survivorship care guidelines, and quality of life (distal outcomes) versus the usual care control arm. In Phase I, community-based participatory research (CBPR) principles will be used to develop the intervention to educate participants about culture and communication by demonstrating how to ask for and verify information with doctors and use personalized symptom reports, and by providing question prompt lists for doctor visits. In Phase II, the intervention will be tested in a pilot randomized control trial (RCT). Using cases from Los Angeles Cancer Surveillance Program, California Cancer Registry, Maryland Cancer Registry, and clinics from California, 118 Chinese immigrant women (diagnosed with stage 0-III breast cancer and 1-3 years post-diagnosis) will be enrolled and randomized to either the E-Talkcare intervention or a usual care control arm. Participants will be interviewed via telephone at baseline (i.e., pre-randomization), 3-, and 6-months post-randomization.

ELIGIBILITY:
Inclusion Criteria:

Eligible Chinese women

* ≥ age 18
* foreign-born speaking Mandarin and/or Cantonese,
* diagnosed with breast cancer at stage 0, I, II or III,
* 1-3 years post-diagnosis and completed primary treatment (surgery, radiation, and chemotherapy); and
* no recurrence, and 6) internet access.

Exclusion Criteria:

* Women with other cancer types are ineligible due to different treatment complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Medical Communication Competence Scale | 6 months
  16 items to assess information provision, seeking, and verifying; α=.80-.89.
Assessment of Patient Experiences of Cancer Care | 6 months
  10-item patient-reported communication quality with follow-up care doctors; α=.75 in Chinese
Decision-making Participation Self-efficacy Scale | 6 months
  5-item measure of patient's efficacy in engaging in medical communication; α=.89 in Chinese
Perceived Personal Control Scale | 6 months
  4-item measure of patients' perceived personal control over breast cancer; α=.71 in Chinese

SECONDARY OUTCOMES:
PROMIS Fatigue | 6 months
  6 items (e.g., felt tired, exhausted, limited at work); α=.97
PROMIS Sleep Disturbance | 6 months
  6 items (e.g., sleep not steady, unsatisfied, hard to fall asleep); α=.98
PROMIS Pain Interference | 6 months
  6 items (e.g., affecting ability to focus, interact with others, run errands); α=.95
PROMIS Cognitive Function | 6 months
  6 items (e.g., had trouble concentrating, slow thinking, hard to concentrate); α=.95
PROMIS Physical Function | 6 months
  8 items (e.g., carry heavy objects, kneeling, doing 2-hour labor work); α=.90
PROMIS Anxiety | 6 months
  7 items (e.g., felt anxious, nervous, fearful, tense); α=.90
PROMIS Depression | 6 months
  8 items (e.g., felt helpless, depressed, unhappy, hopeless); α=.90
Side/late Effect Assessments | 6 months
  31-item measure of patient-reported side/late effects from breast cancer treatment
Adherence to Breast Care Guidelines | 6 months
  26 yes-no items: receiving breast cancer follow-up care recommendations from doctors

CONTACTS AND LOCATIONS:
Overall Officials: Judy Wang, Ph.D., Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT03413332/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT03413332/SAP_001.pdf